CLINICAL TRIAL: NCT04234347
Title: Long Versus Short Axis Approach for Ultrasound Guided Peripheral Intravenous Access: A Randomized Control Trial
Brief Title: Long Versus Short Axis Approach for Ultrasound Guided Peripheral Intravenous Access
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Principal Investigator, Ryan Gibbons, Assistant Professor of Emergency Medicine, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26147
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Venous Access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long Axis approach (Active Comparator): Utilize the longitudinal orientation when placing an USGPIV.
  Interventions: Procedure: Intravenous access method
- Short axis approach (Active Comparator): Utilize the transverse orientation when placing an USGPIV.
  Interventions: Procedure: Intravenous access method

INTERVENTIONS:
Procedure: Intravenous access method — Comparing long and short axis approach to USGPIV access.

SUMMARY:
To compare a long axis approach versus short axis when placing peripheral IVs using ultrasound guidance.

DETAILED DESCRIPTION:
Patients needing an USGPIV will be randomized into long or short axis orientation. Emergency Medicine residents will place the IV using an ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable patients requiring placement of an USGPIV.

Exclusion Criteria:

* Hemodynamically unstable
* Unable to consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
First pass success | 1 day
  USGPIV access
Number of attempts | 1 day
  USGPIV access
Overall success | 1 day
  USGPIV access
Time to completion | 1 day
  USGPIV access

SECONDARY OUTCOMES:
Complications | 1 day
  USGPIV access

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C Gibbons, MD, Principal Investigator — Temple University
Locations (1):
- Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736